CLINICAL TRIAL: NCT01644773
Title: Phase I Study of the Combination of Crizotinib and Dasatinib in Pediatric Research Participants With Diffuse Pontine Glioma (DIPG) and High-Grade Glioma (HGG)
Brief Title: Study of the Combination of Crizotinib and Dasatinib in Pediatric Research Participants With Diffuse Pontine Glioma (DIPG) and High-Grade Glioma (HGG)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJHG12; NCI-2012-01240 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Diffuse Intrinsic Pontine Glioma; High-grade Glioma
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Glioma | interventions — Crizotinib; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Chemotherapy (Experimental): Research participants with high grade glioma or diffuse intrinsic pontine glioma will receive crizotinib and dasatinib.
  Interventions: Drug: Crizotinib; Drug: Dasatinib

INTERVENTIONS:
Drug: Crizotinib — Starting dose level:
  * Initial Treatment Plan: 130 mg/m^2 per dose
  * Modified Treatment Plan per Amendment 1.0: 165 mg/m^2 per dose
  The dose of a single agent will be increased by approximately 30% in each subsequent cohort until the MTD of this combination is reached.
  The doses of each agent will not exceed their single-agent MTD already determined for children with recurrent solid tumors.
  Cycle 1 (28 days): once a day for 28 days
  Cycles 2-26 (28 days each): once a day
  Other Names: PF-02341066; Xalkori®
Drug: Dasatinib — Starting dose level: 50 mg/m^2 per dose
  The dose of a single agent will be increased by approximately 30% in each subsequent cohort until the MTD of this combination is reached.
  The doses of each agent will not exceed their single-agent MTD already determined for children with recurrent solid tumors.
  Cycle 1 (28 days): starting on day 3, once a day for 28 days
  Cycles 2-26 (28 days each): once a day
  Other Names: BMS-354825; Sprycel®

SUMMARY:
This is a phase I study to find the highest tolerable dose of crizotinib and dasatinib given in combination to patients with diffuse intrinsic pontine glioma (DIPG) and other types of high grade gliomas (HGG). Participants will receive escalating doses until the highest dose is determined. Participants will be enrolled in two strata: stratum A for recurrent/ progressive tumors and stratum B for recently diagnosed patients who have completed standard radiation therapy without progressive disease. Up to 7 dosage levels will be tested. Both drugs are taken orally daily, once per day. Correlative pharmacokinetic and biology studies are planned, as well as advanced methods of magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
The Rolling 6 design will be used to estimate the maximum tolerated dose (MTD) and determine the dose-limiting toxicity (DLT) of the combination of escalating doses of crizotinib and dasatinib. Our goal is to accrue research participants for both stratum A and B. However, it is our expectation that the accrual of research participants to stratum B will proceed at a slower pace. Therefore, initially the strategy of dose escalation will be exclusively based on research participants treated at stratum A until the MTD of this combination is reached. Until the MTD of this combination is reached for research participants in stratum A, accrual of research participants in stratum B will be allowed at the highest dosage level which has already been deemed to be safe (i.e., no DLTs in three research participants or ≤ 1 DLT in six research participants). No research participants will be accrued to stratum B until at least one dosage level has been confirmed to be safe in stratum A. Once the MTD for stratum A is reached, we will accrue research participants at this same dosage level to stratum B following the rules of the Rolling 6 design. If the MTD for stratum A is well tolerated among research participants in stratum B, we will proceed with dose escalation for research participants in stratum B based on the same rules of the Rolling 6 design. This strategy is based on the premise that research participants who are more heavily pre-treated (stratum A) may not tolerate therapy as well as those with minimal previous treatment (stratum B).

Primary Objectives:

* To estimate the MTD of the combination of crizotinib (c-Met and ALK inhibitor) and dasatinib (bcr-abl, PDGFRA and B, src, lck, yes, and c-kit inhibitor) in pediatric research participants with recurrent or progressive DIPG and other HGGs (stratum A).
* To estimate the MTD of the combination of crizotinib and dasatinib in research participants with DIPG or HGG who completed RT within a short interval prior to enrollment but have not experienced disease progression (stratum B).

ELIGIBILITY:
Inclusion Criteria: ALL RESEARCH PARTICIPANTS

* Diagnosis of high-grade glioma (HGG) or diffuse intrinsic pontine glioma (DIPG). If histologic confirmation was obtained, diagnosis must be one of the following: anaplastic astrocytoma (WHO grade 3), anaplastic oligodendroglioma (WHO grade 3), anaplastic oligoastrocytoma (WHO grade 3), anaplastic ganglioglioma (WHO grade 3), pleomorphic xanthoastrocytoma with anaplastic features (WHO grade 3), malignant glioneuronal tumor, glioblastoma, or gliosarcoma (WHO grade 4)
* Age > or = 2 years and < or = 21 years
* Performance score > or = 50 (Lansky for research participants < or = 16 years and Karnofsky for those > 16 years).
* Adequate organ function at the time of enrollment as follows:

  * Bone marrow: Hemoglobin > or = 8g/dL [may have received packed red blood cell transfusion], absolute neutrophil count (ANC) > or = 1000/mm^3, platelets > or = 100,000/mm^3 [transfusion independent])
  * Renal: Normal serum creatinine based on age as shown below or GFR > 70ml/min/1.73m^2:

    * Age < or = 5 years: 0.8 mg/dL maximum
    * Age 5 to 10 years: 1.0 mg/dL maximum
    * Age 10 to 15 years: 1.2 mg/dL maximum
    * Age > 15 years: 1.5 mg/dL maximum
  * Hepatic: SGPT and SGOT < 3x the institutional upper limit of normal (ULN), total bilirubin concentration < 1.5x the institutional ULN, albumin > or = 2g/dL
* Female research participants > or = 10 years of age or post-menarchal must not be pregnant (confirmed by serum or urine pregnancy test within 1 week of study enrollment) or breastfeeding
* Female research participants of childbearing age or males research participants of child fathering potential must agree to use safe contraceptive methods for the duration of the study and for 3 months thereafter

Inclusion Criteria: STRATUM A

* Diagnosis of recurrent or progressive HGG or DIPG.
* Neurological deficits must be stable on a fixed or decreasing dose of dexamethasone for ≥7 days before study enrollment.
* Recovery to ≤ grade 1 from all significant toxicities of previous therapies.
* Irradiation: Interval from the last dose of local radiation therapy (RT), craniospinal RT, and palliative RT for symptomatic disease > or = 3 months, > or = 6 months, and > or = 2 weeks before study enrollment, respectively
* Myelosuppressive chemotherapy: Interval > or = 6 weeks and > or = 4 weeks from last dose of nitrosourea and other chemotherapy drugs before study enrollment, respectively. However, interval must be > or = 1 week from last dose of oral etoposide and other drugs administered at low doses (metronomic regimen) before study enrollment
* Small-Molecule Inhibitors: Interval > or = 1 week from last dose before study enrollment. If a previously used agent has a prolonged half-life, the appropriate interval will be determined after consultation with the principal investigator
* Monoclonal Antibodies: Interval > or = 3 half-lives before study enrollment. Such cases will need to be discussed with the principal investigator
* High-Dose Chemotherapy with Stem-Cell Rescue: Interval > or = 3 months before study enrollment
* Cancer Vaccines and Convection-Enhanced Therapies: Interval > or = 1 month before study enrollment
* Growth Factors: Interval > or = 1 week and > or = 2 weeks before study enrollment for standard and long-acting growth factors (e.g., pegfilgrastim), respectively

Inclusion Criteria: STRATUM B

* Completion of local RT with or without concomitant chemotherapy including temozolomide and radiosensitizing agents (e.g., carboplatin, vorinostat) outside the context of a clinical trial. Any agent administered during RT should have a short half-life so that it should already be completely eliminated by the start of this therapy. If other agents were used concurrently with RT, they will need to be discussed with the principal investigator to assess eligibility
* Interval > or = 4 weeks and < or = 8 weeks from the completion of radiochemotherapy

Exclusion Criteria: ALL RESEARCH PARTICIPANTS

* Metastatic disease for stratum B only
* Concomitant use of other anticancer (except for corticosteroids) or experimental agents
* Use of enzyme-inducing anticonvulsants (EIACs). A minimum interval of 10 days between the last dose of EIAC and start of this therapy will be required for research participants who were previously receiving such medications.
* Pregnant or lactating patients
* Research participants with other clinically significant medical disorders that could compromise their ability to tolerate protocol therapy or would interfere with the study procedures or results
* Prior therapy with a PDGFR or c-Met inhibitor
* Original treatment design: Body surface area ≥ 1.8m2on dosage levels 3b, 4, and 5
* Modified treatment design: Body surface area < 0.55 m^2 for all dosage levels

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2012-11-27 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of combination crizotinib and dasatinib in stratum A patients | 6 weeks after start of therapy for last enrolled participant
Maximum tolerated dose of combination crizotinib and dasatinib in stratum B patients | 6 weeks after start of therapy for last enrolled participant

CONTACTS AND LOCATIONS:
Overall Officials: Anna Vinitsky, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Gibson EG, Campagne O, Selvo NS, Gajjar A, Stewart CF. Population pharmacokinetic analysis of crizotinib in children with progressive/recurrent high-grade and diffuse intrinsic pontine gliomas. Cancer Chemother Pharmacol. 2021 Dec;88(6):1009-1020. doi: 10.1007/s00280-021-04357-4. Epub 2021 Sep 29. PMID 34586478
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols